CLINICAL TRIAL: NCT01656967
Title: Flexible Optical Intubation Via the AMBU Aura-I Versus Blind Intubation Via the Fastrach Single Use Intubating LMA - A Prospective Randomized Clinical Trial
Brief Title: AMBU AScope2 Fiberoptic Intubation Versus Fastrach Intubating LMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Ambu A/S (Industry)
Responsible Party: Principal Investigator, Carin A. Hagberg, Professor and Chair, Department of Anesthesiology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-10-0604
Record Dates: First submitted 2012-07-30; First posted 2012-08-03 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Supraglottic Airway
Keywords: Laryngeal Mask Airway; LMA; Intubation; AMBU; AScope; Aura-I; Fastrach; Fiberoptic; Disposable Fiberoptic; Blind Intubation; Fiberoptic Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMBU Aura-I/aScope 2 (Experimental): First, the AMBU Aura-I LMA will be inserted. Then, the patient will be intubated with assistance of the AMBU aScope 2 disposable fiberoptic system.
  Interventions: Device: AMBU Aura-I/aScope 2
- LMA Fastrach (Experimental): The LMA Fastrach Single Use Laryngeal Mask Airway will be placed, followed by blind intubation using the LMA Fastrach EndoTracheal Tube.
  Interventions: Device: LMA Fastrach Single Use

INTERVENTIONS:
Device: AMBU Aura-I/aScope 2 — Once ventilation is achieved, the patients in group A will be intubated through the shaft of Aura-I via the the Ambu aScope.
  Arms: AMBU Aura-I/aScope 2
Device: LMA Fastrach Single Use — The patients in group B will be intubated by ETT via the Intubating LMA as is standard procedure.
  Arms: LMA Fastrach

SUMMARY:
The purpose of this study is to compare two types of supraglottic airways (SGA), the Ambu® Aura-I and the Intubating Laryngeal Mask Airway (ILMA), regarding time to intubate, ease of insertion, sealing properties, optical view upon fiberoptic examination regarding the Ambu Aura-I, ease and success rate of intubation, airway morbidity, and patient comfort in patients undergoing general anesthesia for elective surgery.

DETAILED DESCRIPTION:
The study will include a total of 66 patients. Patients will be randomized into 2 groups through a computer generated randomization schedule. Patients in group A (N= 30) will be intubated using Ambu Aura-I and the Ambu aScope and patients in group B (N= 30) will be intubated using Intubating LMA. Patients will only be tested with one device.In the operating room, standard monitoring devices will be applied including a pulse oximeter, 3 lead (at least) ECG and blood pressure cuff; the latter could be invasive or non-invasive depending on the nature of the surgery. Baseline measures of BP, pulse, oxygen saturation, and CO2 will be made. The time will be noted before any sedation or anesthesia is administered. Vital signs will be recorded after induction of anesthesia, after insertion of SGA, and again after successful intubation.

General anesthesia will be induced by bolus administration of propofol (1.5 to 2mg/kg) and fentanyl (1mcg/kg), and maintained with an inhalational agent. Rocuronium (0.6 mg/kg) will be administered to provide muscle relaxation and a mixture of sevoflurane or isoflurane and nitrous oxide will be utilized for maintenance of anesthesia once the ability to mask ventilate is confirmed. The lungs will be mechanically ventilated with a semi-closed circle system to maintain an end-tidal CO2 near 35 mmHg. Patients' lungs will be ventilated via anesthesia mask 100% oxygen until the patient is completely relaxed.

The size of the SGA device used will be based on manufacturer's recommendations and clinical evaluation of the anesthesiologist. The SGA device will be placed using standard technique and jaw lift will always be performed to aid in placement. The user will record ease of insertion on a scale (1-5) and number of insertions required will also be recorded. A new attempt is considered to begin if the tip of the cuff is withdrawn to the level of the lips. Accurate ventilation is achieved when the CO2 signal is rectangular and the mask is airtight at a respiratory pressure of up to 20 cm H2O. Time will be recorded from when the tip of the device cuff is at the mouth opening and stopped when first CO2 waveform is recorded.

Once ventilation is achieved, the patients in group A will be intubated through the shaft of Aura-I via the the Ambu aScope. If the epiglottis is down folded and obscuring optical view, jaw lift can be performed by an assistant to improve visualization of the cords. The aScope will be advanced until the carina is visualized and then the ETT is railroaded via the aScope into position (5cm above carina or cuff of ETT just below vocal cords). Once the ETT is successfully inserted, the cuff of the Aura-I will be deflated and the patient is ventilated via the ETT. If it is not possible to intubate, the ETT should be rotated 90° counterclockwise and jaw lift should be performed to help with intubation. If unsuccessful after two attempts, the anesthesiologist will proceed to intubate in standard fashion. The patients in group B will be intubated by ETT via the Intubating LMA as is standard procedure.

Once the procedure has finished and the patient is adequately reversed as determined by nerve stimulation, the cuff will be reinflated and the ETT will be removed. Ventilation will resume via the SGA. Once the ETT is withdrawn, the cuff will be adjusted to 60cm H2O using a cuff pressure manometer. The oropharyngeal leak pressure(OLP) is determined with a 60 cm H2O intracuff pressure by closing the expiratory spill valve and then closing the expiratory valve of the circle system at a fixed gas flow of 3 L/min, without any respiration. The airway pressure at which equilibrium is reached and air leaks from the mouth or into the stomach, as sign of leak of the laryngeal mask is noted. Esophageal leak is determined by stethoscopy of the epigastrium and oropharyngeal leak is dectected listening for air leak over the mouth.

The peak airway pressure is not allowed to exceed 40 cmH2O. After OLP measurement and once the patient is adequately breathing on their own, the SGA can be removed.

ELIGIBILITY:
Inclusion Criteria:

* Adult surgical Candidates Aged 18-80 years
* ASA I-III
* Mallampati Score of I or II
* BMI ≤ 35 kg/m2
* Presenting for elective surgery
* Require General Endotracheal Anesthesia.

Exclusion Criteria:

* Previously known difficult airway,
* Emergency status
* Require prone positioning
* Interincisor distance < 2.5cm
* Thyromental distance < 5cm
* Clinically suspected difficult airway
* Contraindications to LMA Insertion, such as Reflux disease
* Patients who do not require endotracheal intubation
* Indications for Rapid Sequence Induction (RSI)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carin A Hagberg, MD, Principal Investigator — The University of Texas Medical School at Houston
Locations (1):
- Memorial Hermann Hospital - Texas Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- AMBU Aura-I/aScope 2: First, the AMBU Aura-I LMA will be inserted. Then, then patient will be intubated with assistance of the AMBU aScope 2 disposable fiberoptic system.
  AMBU Aura-I LMA and aScope 2 Disposable Fiberoptic Camera
- LMA Fastrach: The LMA Fastrach Single Use Laryngeal Mask Airway (The Laryngeal Mask Airway Company, California) will be placed, followed by blind intubation using the LMA Fastrach EndoTracheal Tube.
  LMA Fastrach Single Use
Period: Overall Study
Arm/Group | AMBU Aura-I/aScope 2 | LMA Fastrach
Started | 33 | 33
SGA Placement | 32 | 33
ETT Insertion | 29 | 31
Completed | 29 | 31
Not Completed | 4 | 2
Not completed — faulty monitor | 1 | 0
Not completed — unsuccessful ETT insertion | 3 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled patients, except for one in the Ambu group who was withdrawn due to a faulty monitor
Groups:
- Total: Total of all reporting groups
Arm/Group | AMBU Aura-I/aScope 2 | LMA Fastrach | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (13.7) | 44.4 (13.7) | 42.1 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 20 | 18 | 38
Region of Enrollment [Number; unit: participants]
  United States | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: Total Intubation Time
Description: Total Intubation Time includes time for SGA insertion and for ETT insertion. The total time to intubation was measured from the beginning of SGA insertion to successful endotracheal tube intubation verified by detection of CO2 on the capnogram.
Time Frame: Duration of Intubation, including supraglottic airway (SGA) insertion and endotracheal tube (ETT) insertion
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | AMBU Aura-I/aScope 2 | LMA Fastrach
Number analyzed (Participants) | 29 | 31
seconds | 89.6 [67.8 to 117.5] | 52.1 [46.4 to 69.8]

2. Secondary Outcome: Time for Supraglottic Airway (SGA) Insertion
Description: Time for SGA insertion was measured from when the tip of the cuff was at the mouth to detection of CO2 on the capnogram.
Time Frame: At SGA insertion
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | AMBU Aura-I/aScope 2 | LMA Fastrach
Number analyzed (Participants) | 32 | 33
seconds | 28.6 [20.9 to 37.9] | 30.3 [23.0 to 36.8]

3. Secondary Outcome: Time for Endotracheal Tube (ETT) Insertion
Description: After the SGA is inserted, time for intubation will be recorded. Time for ETT insertion was measured, for arm 1, from when the AMBU aScope is at the connector level of the Aura-I or, for arm 2, from when the ETT is at the connector level of the Intubating LMA to first detection of CO2 on the capnogram. The AScope 2 disposable fiberoptic camera will be used to assist with intubation for Group 1 patients. Group 2 patients will be intubated using the LMA-Fastrach EndoTracheal Tube.
Time Frame: At ETT insertion
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | AMBU Aura-I/aScope 2 | LMA Fastrach
Number analyzed (Participants) | 29 | 31
seconds | 60.9 [41.0 to 84.0] | 23.1 [20.6 to 33.0]

4. Secondary Outcome: Number of Participants in Whom SGA Insertion Was Successful on the First Attempt
Time Frame: At SGA insertion
Measure: Number; unit: participants
Arm/Group | AMBU Aura-I/aScope 2 | LMA Fastrach
Number analyzed (Participants) | 32 | 33
participants | 30 | 30

5. Secondary Outcome: Number of Participants in Whom ETT Insertion Was Successful on the First Attempt
Time Frame: At ETT insertion
Measure: Number; unit: participants
Arm/Group | AMBU Aura-I/aScope 2 | LMA Fastrach
Number analyzed (Participants) | 32 | 33
participants | 26 | 27

6. Secondary Outcome: Number of Participants With Overall Success for SGA Placement
Description: Ease of SGA insertion is subjectively assessed by the operator on a scale from 1 to 5 (1 = extremely easy, 5 = extremely difficult).
Time Frame: At SGA insertion
Measure: Number; unit: participants
Groups:
- AMBU Aura-I/aScope 2: First, the AMBU Aura-I LMA will be inserted. Then, then patient will be intubated with assistance of the AMBU aScope 2 disposable fiberoptic system.
  AMBU Aura-I LMA and aScope 2 Disposable Fiberoptic Camera
  first-attempt success rate for SGA placement for the Aura-i group (30/33, 90.9%)
- LMA Fastrach: The LMA Fastrach Single Use Laryngeal Mask Airway (The Laryngeal Mask Airway Company, California) will be placed, followed by blind intubation using the LMA Fastrach EndoTracheal Tube.
  LMA Fastrach Single Use
  first-attempt success rate for SGA placement for the ILMA group (30/33, 90.9%, P = 1.0)
Arm/Group | AMBU Aura-I/aScope 2 | LMA Fastrach
Number analyzed (Participants) | 33 | 33
participants | 30 | 30

7. Secondary Outcome: Number of Participant With Overall Intubation Success
Description: Ease of ETT insertion is subjectively assessed by the operator on a scale from 1 to 5 (1 = extremely easy, 5 = extremely difficult).
Time Frame: At ETT insertion
Measure: Number; unit: participant
Arm/Group | AMBU Aura-I/aScope 2 | LMA Fastrach
Number analyzed (Participants) | 33 | 33
participant | 29 | 31

8. Secondary Outcome: Post-Operative Discomfort Upon Entering the Post-Anesthesia Care Unit (PACU)
Description: The patient will be assessed for Post-Operative Hoarseness, Sore Mouth, Sore Neck, Sore Jaw, Dysphonia, Dysphagia, and Altered Tongue Sensation.
Time Frame: Within 30 minutes of completion of surgery
Measure: Number; unit: participants
Arm/Group | AMBU Aura-I/aScope 2 | LMA Fastrach
Number analyzed (Participants) | 33 | 33
participants | 29 | 30

9. Secondary Outcome: Post-Operative Discomfort Upon Leaving the Post-Anesthesia Care Unit (PACU)
Description: as for outcome 8
Time Frame: Approximately 1-2 hours after entering the PACU
Measure: Number; unit: participants
Arm/Group | AMBU Aura-I/aScope 2 | LMA Fastrach
Number analyzed (Participants) | 33 | 33
participants | 29 | 30

10. Other Pre Specified Outcome: Orolaryngeal Pressure
Description: The oropharyngeal leak pressure (OLP) was determined by closing the expiratory valve of the circle system at a fixed gas flow of 3 L/min and noting the airway pressure at which equilibrium was reached (not permitted to exceed 40 cm H2O).
Time Frame: Following SGA Insertion
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | AMBU Aura-I/aScope 2 | LMA Fastrach
Number analyzed (Participants) | 32 | 33
mmHg | 28.0 [24.5 to 30.0] | 26.0 [24.0 to 30.0]

ADVERSE EVENTS:
Time Frame: Adverse Event data include measures of post-operative discomfort upon entering the Post-Anesthesia Care Unit (PACU). Patients entered the PACU within 30 minutes of completion of surgery. Data collected for 6 months duration.
Arm/Group | AMBU Aura-I/aScope 2 | LMA Fastrach
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 3/29 | 8/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMBU Aura-I/aScope 2 (N=29) | LMA Fastrach (N=31)
Hoarseness (Surgical and medical procedures) | 1 (13) | 2 (16)
Sore mouth (Surgical and medical procedures) | 3 (29) | 8 (31)
Sore neck (Surgical and medical procedures) | 1 (1) | 3 (3)
Sore Jaw (Surgical and medical procedures) | 0 (0) | 1 (1)
Dysphonia (Surgical and medical procedures) | 1 (5) | 1 (7)
Dysphagia (Surgical and medical procedures) | 3 (21) | 2 (22)
Altered tongue sensation (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Experience of the residents, some only had 6 months experience When using AScope, there were secretions and no suctioning capability Sample size ILMA is a straightforward attempt; whereas, AScope needs to maneuver and go all the way to carina

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No